CLINICAL TRIAL: NCT00738413
Title: An Iron Balance Study Comparing Deferasirox, Deferoxamine and the Combination of Both Drugs
Brief Title: Iron Balance Study of Deferasirox, Deferoxamine and the Combination of Both
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Robert W. Grady, Ph.D., Weill Cornell Medical College
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0804009771; DK55463
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2010-11

CONDITIONS: Thalassemia
Keywords: Iron chelation; Iron balance; Secondary iron overload; deferoxamine; deferasirox
MeSH Terms: conditions — Thalassemia | interventions — Deferoxamine; Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Active Comparator): Subjects will be treated for 6 days with deferoxamine.
  Interventions: Drug: Deferoxamine
- Arm 2 (Active Comparator): Subjects will be treated for 6 days with deferasirox.
  Interventions: Drug: Deferasirox
- Arm 3 (Experimental): Subjects will be treated for 6 days with a combination of deferoxamine and deferasirox.
  Interventions: Drug: Deferoxamine; Drug: Deferasirox

INTERVENTIONS:
Drug: Deferoxamine — Deferoxamine will be administered subcutaneously over 8 hours for 6 days at a dose of 40 mg/kg.
  Other Names: Desferal, DFO
  Arms: Arm 1; Arm 3
Drug: Deferasirox — Deferasirox will be orally administered at a dose of 30 mg/kg once daily for 6 days.
  Other Names: Exjade, ICL670
  Arms: Arm 2; Arm 3

SUMMARY:
Subjects with thalassemia major require regular transfusion therapy to sustain life. The iron present in the transfused blood remains in the body where it can cause a variety of organ dysfunctions. Lifelong iron chelation therapy is needed to maintain iron balance but its effectiveness varies greatly. Like that of deferoxamine (Desferal, DFO) the mainstay of chelation therapy for 30 years, the effectiveness of deferasirox (Exjade, ICL670), the newly approved, orally effective iron chelating drug, is not satisfactory in all subjects. Even with good compliance, the iron excretion induced by a given drug exhibits wide subject-to-subject variability. There is often persistent iron overload of extra hepatic tissues such as the heart and pancreas leading to cardiac disease and diabetes. Combining the drugs may be a better approach in those subjects at increased risk. The iron balance studies proposed will permit an assessment of the potential of such a combination to place subjects in net negative iron balance and the relative effectiveness of the combination in relation to that of the individual drugs, an additive effect being expected. With such information, physicians will be able to design individualized chelation regimens that maximize effectiveness while minimizing side effects by adjusting the ratio and/or the dosing schedule of the two drugs.

DETAILED DESCRIPTION:
The study involves a 34-day hospital stay during which we will conduct metabolic iron balance studies wherein deferasirox and deferoxamine are evaluated separately and in combination, each subject serving as his/her own control. In the studies currently proposed, deferasirox (20, 30 or 40 mg/kg, administered p.o. 30 minutes before breakfast) and deferoxamine (30, 40, 50 or 60 mg/kg infused subcutaneously over 8 hours at night) will be evaluated both alone and in combination, the drugs being given sequentially as above or simultaneously wherein deferasirox is administered 30 minutes after beginning the infusion of deferoxamine. In the first phase of the studies, the combination of drugs will be given sequentially, deferasirox 30 minutes prior to breakfast at a dose of 30 mg/kg and deferoxamine during the night at 40 mg/kg.

On days 5 - 10, the subjects will receive their first chelation regimen, deferoxamine infused subcutaneously over 8 hours during the night. They will receive a daily multivitamin preparation containing 60 -100 mg of vitamin C, 1 mg of folic acid and 400 I.U. of vitamin E. On days 15 - 20, the subjects will be given deferasirox 30 minutes prior to breakfast. Finally, on days 25 - 30, the subjects will receive both deferoxamine and deferasirox, the combination of drugs being given either sequentially (deferasirox in the morning and deferoxamine at night) or simultaneously (infusion of deferoxamine beginning 30 minutes prior to taking deferasirox). Non-drug days allow for clearance of stool iron induced by the previous treatment. A period of 4 days was chosen because this includes the normal gastrointestinal transit time of most individuals. A stool marker (brilliant blue) will be administered before the first and after the last dose of each drug to help in quantifying fecal iron excretion.

Upon admission and discharge, each subject will be given a complete physical examination and various clinical and laboratory parameters will be measured. These include a routine blood profile (complete blood count with differential, and platelet count), a serum chemistry profile (fasting blood sugar, total protein, albumin, AST, ALT, BUN, creatinine, bilirubin (total), bilirubin (direct), alkaline phosphatase, uric acid, calcium, phosphorus, magnesium, zinc, copper, sodium, potassium, chloride and carbon dioxide) and a urinalysis (protein, beta-2 microglobulin, glucose, ketones, hemoglobin, pH, specific gravity and bacteria; if abnormal, a microscopic examination for RBC, WBC, casts, crystals and cells). Additional blood tests to be done at admission include serum ferritin, serum iron, iron binding capacity, % saturation, vitamin C, a serum pregnancy test, hepatitis C antibody and HIV-PCR with viral load. At the beginning and end of the study, an ophthalmology workup including a slit lamp and retinal examination, an audiogram, and an electrocardiogram will also be performed. In addition to those studies conducted upon admission and discharge, serial blood tests and urinalyses will be done on days 6, 10, 14, 16, 20, 24, 26 and 30 to ensure adequate monitoring of organ function.

Each subject will be placed on a fixed low-iron diet consisting of four rotating meal plans designed by our nutritionists in consultation with the subjects themselves. Twenty-four hour specimens of urine and stool will be collected daily and their iron content determined by atomic absorption. Net excretion will be determined taking into account the iron content of all uneaten food. The excretion of copper and zinc will also be monitored to insure that these physiologically important metals are not depleted. Each subject will be given a unit of blood on days 1, 11, 21 and 34. This will ensure that the level of erythropoiesis is approximately the same before each drug regimen.

In order to reduce the stress and boredom of the 34-day hospitalization, it is anticipated that the subjects will be studied in pairs so that they will always have someone in a similar situation to interact with. They will have free access to television, the internet and local phone service while in the clinical research unit. The subjects must eat breakfast and dinner in the research unit and sleep there. Otherwise, they may go out on pass during the day and after dinner in the evenings for shopping, entertainment, etc. We will pack their lunch if they choose to go out for the day as they will not be allowed to consume any food or drink other than what is provided in their agreed upon diet. Visitors will be allowed during normal hospital visiting hours.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with transfusional iron overload secondary to thalassemia major, aged 18 or older, may participate after giving written informed consent. Subjects must have no clinically significant finding in their medical history, on physical examination or as a result of laboratory assessments other than those consistent with thalassemia major and its complications, such as compensated cirrhosis, endocrine insufficiency and diabetes.
* Subjects must have a serum ferritin greater than 1000 ng/mL, a platelet count greater than 100,000/mm3, and a serum creatinine within the normal range.
* Subjects must be willing and able to discontinue their usual regimen of DFO, deferiprone (L1, Ferriprox) or Exjade for the duration of the study.
* A woman of childbearing potential must have a negative serum pregnancy test at screening. She must use a medically acceptable form of birth control during the study and for 1 month afterward. Acceptable birth control measures include: abstinence, oral contraceptives, hormonal contraceptive implants, barrier contraceptives (condom, diaphragm with spermicide), IUD, and/or a vasectomized partner. Male subjects must also use barrier contraceptives during the study and for 1 month thereafter.
* The subjects must also have a level of understanding and willingness to cooperate with the confinement and procedures described in the consent form and scheduled by the study site. In addition, he/she must be able to provide voluntary written informed consent.
* Subjects must weigh at least 40 kg.

Exclusion Criteria:

* Subjects can not have a history of clinically significant gastrointestinal, renal, hepatic, endocrine, oncologic, infectious, pulmonary or cardiovascular disease, other than conditions associated with thalassemia and iron overload, such as compensated cirrhosis, endocrine insufficiency and diabetes, or a history of tuberculosis, epilepsy, psychosis, glaucoma or any other condition, which in the opinion of the investigators, would jeopardize the safety of the subject or impact the validity of the study results.
* Subjects can not be HIV positive or have active HCV.
* A history of serious immunologic hypersensitivity to any medication, such as anaphylaxis or angioedema.
* Participation in a previous investigational drug study within the 30 days preceding screening. A chelation regimen including deferiprone or Exjade within 30 days of screening would not exclude subjects coming from regions where these drugs are an approved medication.
* Women who are pregnant, or breast-feeding.
* Current alcohol or drug abuse.
* An inability to adhere to the designated procedures and restrictions of this protocol.
* Subjects with abnormal or irregular bowel function (defined as more than 3 bowel movements/day or less than 1 bowel movement every other day).
* Subjects receiving warfarin, digoxin, or anti-arrhythmic or anti-seizure medications.
* Subjects with a known allergy to Exjade or DFO that prevents chronic administration.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-09 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is to assess the safety and tolerability of combining DFO and deferasirox in thalassemia subjects with translation iron overload. | 34 days

SECONDARY OUTCOMES:
The secondary outcome measure is to determine the relative level of iron balance achieved upon administering the drugs in combination compared to that upon giving the drugs individually. | 34 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Grady, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Grady RW, Galanello R, Randolph RE, Kleinert DA, Dessi C, Giardina PJ. Toward optimizing the use of deferasirox: potential benefits of combined use with deferoxamine. Haematologica. 2013 Jan;98(1):129-35. doi: 10.3324/haematol.2012.070607. Epub 2012 Aug 8. PMID 22875626